CLINICAL TRIAL: NCT04629378
Title: A Phase 2 Trial to Evaluate the Early Bactericidal Activity and Safety of Meropenem With Amoxicillin/Clavulanate Plus Either Pyrazinamde or Bedaquiline in Adults With Newly Diagnosed Rifampicin-susceptible Pulmonary Tuberculosis
Brief Title: Evaluating the EBA of Meropenem With Amoxicillin/Clavulanate and Pyrazinamide or Bedaquiline in Adults With PTB
Acronym: TB_COMBO_01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TASK Applied Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASK-005_TB_COMBO_01
Record Dates: First submitted 2020-10-12; First posted 2020-11-16 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2020-11

CONDITIONS: Tuberculosis
Keywords: tuberculosis; TB; early bactericidal activity
MeSH Terms: conditions — Tuberculosis | interventions — Meropenem; Amoxicillin-Potassium Clavulanate Combination; Pyrazinamide; bedaquiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Meropenem and amoxicillin/clavulanate plus pyrazinamide (Experimental): Meropenem administered intravenously once daily over 6 hours plus amoxicillin/clavulanate 2 x 1000/62.5 mg once daily orally plus pyrazinamide 20-30 mg/kg orally once daily. All study treatments will be administered for 14 consecutive days.
  Interventions: Drug: Meropenem Injection; Drug: Amoxicillin Clavulanate; Drug: Pyrazinamide
- Meropenem and amoxicillin/clavulanate plus bedaquiline (Experimental): Meropenem administered intravenously once daily over 6 hours plus amoxicillin/clavulanate 2 x 1000/62.5 mg once daily orally plus bedaquiline 400 mg orally once daily. All study treatments will be administered for 14 consecutive days.
  Interventions: Drug: Meropenem Injection; Drug: Amoxicillin Clavulanate; Drug: Bedaquiline
- Rifafour standard of care treatment (Active Comparator): Rifafour e275® administered orally once daily for 14 consecutive days. Rifafour e275® will be administered according to the South African National TB Treatment Guidelines. The daily dose is dependent on the participants' weight as follows: 40 - 54kg: 3 tablets; 55 - 70kg: 4 tablets; 71kg and over: 5 tablets.
  Interventions: Drug: Rifafour

INTERVENTIONS:
Drug: Meropenem Injection — Meropenem IV 6 grams
  Arms: Meropenem and amoxicillin/clavulanate plus bedaquiline; Meropenem and amoxicillin/clavulanate plus pyrazinamide
Drug: Amoxicillin Clavulanate — Amx/CA oral 1000/62.5mg 2 tablets
  Arms: Meropenem and amoxicillin/clavulanate plus bedaquiline; Meropenem and amoxicillin/clavulanate plus pyrazinamide
Drug: Pyrazinamide — Pyrazinamide 20-30mg/kg
  Arms: Meropenem and amoxicillin/clavulanate plus pyrazinamide
Drug: Bedaquiline — Bedaquiline 400mg
  Arms: Meropenem and amoxicillin/clavulanate plus bedaquiline
Drug: Rifafour — Rifafour (HRZE) Standard dose
  Arms: Rifafour standard of care treatment

SUMMARY:
A single-center, open-label clinical trial to determine the early bactericidal activity (EBA) and safety of the combination of meropenem and amoxicillin/clavulanate plus pyrazinamide vs. meropenem and amoxicillin/clavulanate plus bedaquiline administered for 14 consecutive days. This study forms part of a series of 2-week EBA studies to determine the relative bactericidal activity of several new or repurposed anti-tuberculosis agents from which to determine the most effective and safe combination to evaluate in larger and longer duration regimen-based trials.

DETAILED DESCRIPTION:
Study design

A single-center, open-label clinical trial. Study treatments include:

1. Meropenem 6g intravenously once daily plus amoxicillin/clavulante 2 x 1000mg/62.5mg orally once daily and pyrazinamide 20-30mg/kg orally once daily on days 1-14. Ten participants will be included in this treatment arm.
2. Meropenem 6g intravenously once daily plus amoxicillin/clavulanate 2 x 1000mg/62.5mg orally once daily and bedaquiline 400mg orally once daily on days 1-14. Ten participants will be included in this treatment arm.
3. Rifafour e- 275® (HRZE) orally once daily on days 1-14, with weight-banded dosing. Two participants will receive standard first line TB treatment as per the South African TB guidelines (Rifafour e- 275®) and is included as a control for the EBA quantitative mycobacteriology and to evaluate whether HRZE gives similar EBA results to that demonstrated in prior studies with this combination.

Patient Population:

A total of 22 male and female participants aged between 18 and 65 years (inclusive), with newly diagnosed, smear-positive, pulmonary TB will be included.

Treatment

The Investigational Product (IP) will be supplied as:

* Meropenem 1g reconstitution vials
* Amoxicillin/CA 1000/62.5mg tablets
* Pyrazinamide 500mg tablets
* Bedaquiline 100mg tablets

Statistical Methods:

This is a descriptive study with no inferential statistics or hypothesis testing. The planned sample size of 10 participants per treatment group is in keeping with other phase 2 trials of this type and accounts for the possibility of up to 3 drop-outs per arm, which based on previous studies of this type conducted at these sites, represents a conservative estimate of the expected drop-out rate.

Trial Duration:

37 days (up to 9 days pre-treatment plus 15 days treatment period plus 14 days post- treatment follow- up).

ELIGIBILITY:
Inclusion Criteria:

* Provide written, informed consent prior to all trial-related procedures including HIV testing.
* Male or female, aged between 18 and 65 years, inclusive.
* Body weight (in light clothing and with no shoes) between 40 and 90 kg, inclusive.
* Newly diagnosed, previously untreated, rifampicin-susceptible pulmonary TB.
* A chest X-ray picture which in the opinion of the Investigator is consistent with TB.
* Sputum positive on microscopy for acid-fast bacilli on at least one sputum sample (at least 1+ on the IUATLD/WHO scale).
* Ability to produce an adequate volume of sputum as estimated from an overnight sputum collection sample (estimated 10 ml or more).
* Be of non-childbearing potential or using effective methods of birth control throughout participation in the study until Visit 19 (day 28).

Non-childbearing potential:

1. Female participant/sexual partner - bilateral oophorectomy, bilateral tubal ligation and/or hysterectomy or hasbeen postmenopausal with a history of no menses for at least 12 consecutive months; or
2. Male participant/sexual partner - vasectomised or has had a bilateral orchidectomy minimally three month prior to screening;

Effective birth control methods:

1. Participant - not heterosexually active or practicing sexual abstinence; or
2. Double barrier method which can include a male condom, diaphragm, cervical cap, or female condom (male and female condoms should not be used together); or
3. Barrier method combined with hormone-based contraceptives or an intra-uterine device for the female partner.

Exclusion Criteria:

* Evidence of clinically significant conditions or findings, other than the indication being studied, particularly epilepsy, that might compromise safety or the interpretation of trial endpoints, per discretion of the Investigator.
* Poor general condition where any delay in treatment cannot be tolerated per discretion of the Investigator.
* Clinically significant evidence of extrathoracic TB (miliary TB, abdominal TB, urogenital TB, osteoarthritic TB, TB meningitis), as judged by the Investigator.
* Significant history of cardiovascular disease such as heart failure, a personal or family history of congenital QT prolongation, Torsade de Pointes, or QTcF interval > 500 ms (confirmed by repeat electrocardiogram).
* History of allergy to any of the trial IP/s or related substances i.e. β-lactams and penicillin, as confirmed by the clinical judgement of the Investigator.
* Alcohol or drug abuse, that in the opinion of the Investigator, is sufficient to compromise the safety or cooperation of the participant.
* HIV positive ONLY IF:

  * CD4 < 350cells/mm3
  * On ART
* Having participated in other clinical studies with investigational agents within 8 weeks prior to trial start.
* Female participant who is pregnant, breast-feeding, or planning to conceive a child within the anticipated period of participating in the trial. Male participant planning to conceive a child within the anticipated period of participating in the trial.
* Subjects with diabetes (Type 1 or 2), or random glucose over 11.1 mmol/L.
* Hypersensitivity to local anaesthesia of amide type.
* Treatment received with any drug active against Mtb (including but not limited to isoniazid, ethambutol, amikacin, cycloserine, fluoroquinolones, rifabutin, rifampicin, streptomycin, kanamycin, para-aminosalicylic acid, rifapentine, pyrazinamide, thioacetazone, capreomycin, thioamides, metronidazole), or with immunosuppressive medications such as TNF-alpha inhibitors or systemic corticosteroids, within 2 weeks prior to screening.
* Participants with the following toxicities at screening as defined by the enhanced CTCEA toxicity table

  1. creatinine >1.5 times upper limit of normal (ULN);
  2. haemoglobin <8.0 g/dL;
  3. platelets equal to or <50x10E9 cells/L);
  4. serum potassium <3.0 mEq/L;
  5. aspartate aminotransferase (AST) ≥3.0 x ULN;
  6. alanine aminotransferase (ALT) ≥3.0 x ULN;
  7. APTT grade 3
  8. INR grade 3
  9. Total white cell count grade 3

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Early bactericidal activity (EBA) over 14 treatment days based on the rate of change in colony forming unit (CFU) count per treatment arm | 14 days
  CFU count will be determined from Mycobacterium tuberculosis (M.tb) grown on solid culture. The rate of change in CFU count per ml sputum will be determined from overnight sputum samples collected for at least 2 day before study treatment till day 4 on treatment, followed by alternate days till day 14 on treatment.

SECONDARY OUTCOMES:
EBA over 14 treatment days based on the rate of change in time to positive culture (TTP) per treatment arm | 14 days
  TTP will be determined from M.tb grown in liquid culture media. The rate of change in TTP per ml sputum will be determined from overnight sputum samples collected for at least 2 day before study treatment till day 4 on treatment, followed by alternate days till day 14 on treatment.
Safety and tolerability of study treatments administered over 14 consecutive days | 14 days
  Incidence of treatment emergent adverse events (TEAEs) will be summarised by severity, relatedness to study treatments, and seriousness, leading to early withdrawal and/or leading to death, and summarised per treatment arm.
Cmax: Maximum observed plasma drug concentration. | 14 days
  The maximum observed plasma concentration (Cmax), will be estimated for all analytes in all treatment arm, excluding the standard of care arm. Parameter will be calculated separately using plasma concentrations.
Tmax: Time at which Cmax is observed (obtained without interpolation).(interventional arms only) after 14 consecutive days - Analyte, Meropenem; amoxicillin; CA; bedaquiline | 14 days
  The time to reach Cmax (Tmax), will be estimated for all analytes in all treatment arm, excluding the standard of care arm. Parameter will be calculated separately using plasma concentrations.
Cmin: Minimum observed plasma drug concentration 24 hours following the last dose. | 14 days
  The minimum observed plasma concentration (Cmin) 24 hours following intake of the first daily dosing on day 14, will be estimated for all analytes in all treatment arm, excluding the standard of care arm. Parameter will be calculated separately using plasma concentrations.
AUC(0-24): Area under the drug concentration-time curve calculated using linear trapezoidal summation from time zero to time 24 hours. | 14 days
  The 24 hours following intake of the first daily dosing on day 14, area under the plasma concentration time curve from zero to 24 hours (AUC(0- 24)) will be estimated for all analytes in all treatment arm, excluding the standard of care arm. Parameter will be calculated separately using plasma concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Veronique R De Jager, MBChB, Principal Investigator — TASK
Locations (1):
- TASK Clinical Research Centre, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Still in planning.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available once all study activities and publications are finalized and will be made available for the maximum time for which it is still clinically relevant.
Access Criteria: Still in planning.